CLINICAL TRIAL: NCT06230419
Title: Evaluation of Artificial Intelligence's Ability to Analyze and Recognize Cranial Trauma CT Imaging
Brief Title: Retrospective Study on the Direction of Artificial Intelligence in Identifying Cranial Trauma CT Imaging
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Junfeng Feng, Director of Brain Injury Center, RenJi Hospital
Other Study IDs: 83760142
Record Dates: First submitted 2024-01-08; First posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Cerebral Hemorrhage
Keywords: Artificial Intelligence; Computed Tomography
MeSH Terms: conditions — Cerebral Hemorrhage

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- The cerebral trauma group

SUMMARY:
The goal of this observational retrospective study is to evaluate artificial intelligences (AI)'s proficiency in identifying and annotating brain bleeds in computed tomography (CT) images.

The main questions it aims to answer are:

* Whether AIs at present are capable of analyzing and recognizing cerebral traumas in CT images?
* If they are, how competent are they and how can humans take advantages of that? CT images were selected during the normal diagnosis and treatment process of patients, and no one needed to undergo any additional procedures connected to the study.

ELIGIBILITY:
Inclusion Criteria:

* People who had cerebral traumas with brain bleedings shown in CT images.

Exclusion Criteria:

* Brain bleedings were not clear or representative in CT images.

Ages: 16 Years to 92 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population ranges from 16 years old to 92 years old, both female and male, who mostly are the elderly.
Sampling Method: Probability Sample
Enrollment: 208 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-02-15 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
The identification completeness of the annotated images. | 1 months
  Use Photoshop to calculate the area of hemorrhage and the marked area, and then computing the ratio, import into Graphpad Prism for further analysis of the mean percentage and the standard deviation.

SECONDARY OUTCOMES:
The evaluations from professionals for outcomes produced by AIs | 1 months
  The outputs will be evaluated by professional radiologists on a 4-point scale questionnaire from the completeness, accuracy and success of the annotation. Then the results of the questionnaire will be further analyzed in the Graphpad Prism to get the average score and the standard deviation.

CONTACTS AND LOCATIONS:
Locations (1):
- Brain Injury Center, Renji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Zhang D, Ma Z, Gong R, Lian L, Li Y, He Z, Han Y, Hui J, Huang J, Jiang J, Weng W, Feng J. Using Natural Language Processing (GPT-4) for Computed Tomography Image Analysis of Cerebral Hemorrhages in Radiology: Retrospective Analysis. J Med Internet Res. 2024 Sep 26;26:e58741. doi: 10.2196/58741. PMID 39326037